CLINICAL TRIAL: NCT04936204
Title: A Prospective, Randomized, Controlled, Single-blind Clinical Investigation to Evaluate the Safety and Performance of ConnettivinaBio Plus Cream Compared to ConnettivinaBio Cream in the Management of Wounds in Patients at High Risk of Infection
Brief Title: Clinical Investigation to Evaluate the Safety and Performance of ConnettivinaBio Plus Cream Compared to ConnettivinaBio Cream in the Management of Wounds in Patients at High Risk of Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HQQ2-19-01
Record Dates: First submitted 2020-10-07; First posted 2021-06-23 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, single-blind clinical investigation
Who Masked: Outcomes Assessor
Masking Description: At Screening/Baseline visit patients who signed the informed consent and are eligible for the study will be screened by the Investigator who will gather demographic and medical history data and perform the randomization procedure. After the allocation of the patient to Group 1 or 2, the Un-blinded Investigator will perform the treatment, according to the group allocation and instruct the patients on dressing daily renewal. The Investigator, who won't take part in the administration of study treatments and won't be aware on the patient.s group assignment, will perform all the evaluations for primary and secondary endpoint, during the visits (Blinded Evaluator).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 ConnettivinaBio Plus cream (Experimental): ConnettivinaBio Plus cream is a topical preparation constituted by Principal component: Hyaluronic acid sodium salt 0.2% Other components: Silver Sulfadiazine 1%, The medication should be applied once a day as a thin layer to cover the entire surface of the wound previously cleansed
  Interventions: Device: ConnettivinaBio Plus cream
- Group 2 ConnettivinaBio cream (Active Comparator): ConnettivinaBio Cream is a topical preparation constituted by Principal component: Hyaluronic acid sodium salt 0.2% The medication should be applied once a day as a thin layer to cover the entire surface of the wound previously cleansed
  Interventions: Device: ConnettivinaBio cream

INTERVENTIONS:
Device: ConnettivinaBio Plus cream — The Un-blinded Investigator will perform the first application of medication. He will also instruct the patient or his/her caregiver to the self-application of the treatment which will be covered by a secondary dressing according to the site's standard care.
  Other Names: Bionect Plus; Hyalo4 Control
  Arms: Group 1 ConnettivinaBio Plus cream
Device: ConnettivinaBio cream — The Un-blinded Investigator will perform the first application of medication. He will also instruct the patient or his/her caregiver to the self-application of the treatment which will be covered by a secondary dressing according to the site's standard care.
  Other Names: Bionect; Hyalo4 skin
  Arms: Group 2 ConnettivinaBio cream

SUMMARY:
The clinical investigation plan will include a Screening/Baseline visit (V1) in which patients will be screened on the basis of inclusion/exclusion criteria and clinically evaluated. Screened and eligible patients will be randomly assigned in one of the two groups: Group 1 will receive ConnettivinaBio Plus cream whereas Group 2 will receive ConnettivinaBio cream. Lesions will be cleaned and a photo will be acquired with a digital camera.

In both groups, the schedule treatment will consist of daily medication changes.

Wound Bed Score, clinical signs of localized infection, measurement of the wound area, collection of the swab, according to the Levine's technique, EQ-5D questionnaire to the patient will be assessed on Day 1 (V1, baseline visit), 7 (V2), 14 (V3), 21 (V4) and 28 (V5) post-baseline. Treatments in both groups (ConnettivinaBio Plus or ConnettivinaBio) will be applied for a maximum period of 28 days. The easiness of treatment application will be also recorded at V5.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female ≥ 18 years
* Having wounds (both chronic or acute wounds regardless of etiology), with the following characteristics:
* Non infected
* Wound Bed Score ≥4 and <13
* Wound area ≤ 100 cm2
* Patient having one or more factors associated with increased risk of wound infection (IWII, 2016)
* Patient able to read and understand the language and content of the study material, understand the requirements for follow-up visits, is willing to provide information at the scheduled evaluations and is willing, able and ensuring to comply with the study requirements for the whole study period.

Exclusion Criteria:

* Absence of factors associated with increased risk of wound infection
* Infected wounds - where infection is defined by:

For chronic wounds:

A combination of three or more signs or symptoms of local infection: periwound skin erythema, local heat, persistent pain, oedema of wound.s edge, malodour, pus and heavy exudation (Cutting KF, 1994; Trial C, 2010);

For acute wounds:

Cellulitis or pus or abscess, Delayed healing, erythema, hardening of edge, serous-purulent drainage, malodour

* Non-vital tissue greater than 25% of the total wound area
* Heavily exuding wounds
* Presence of fistula
* History of connective tissue disease, e.g., systemic lupus erythematosus, systemic sclerosis, Sjögren's syndrome or mixed connective tissue disease
* Active malignant disease
* Active sickle cell disease
* radiation therapy
* Known allergy to any of the devices' constituents
* Pregnant and breastfeeding women
* Subjects unable to understand informed consent or having a high probability of non- compliance with the study procedures and or non-completion of the study according to investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
improving the wounds bed conditions in wounds at high risk of infection, after 14 days of treatment, compared to ConnettivinaBio cream | at day 14
  The amelioration of wound's bed conditions will be evaluated by measuring the proportion of patients having an increase of at least one subclass of the Wound Bed Score (WBS) (0-16 score; 0 worse score-16 best score possible) (Falanga V, 2006) from baseline to 14 days of treatment with ConnettivinaBio Plus cream compared to ConnettivinaBio cream.

SECONDARY OUTCOMES:
improving the wound bed condition | At days 7, 21 and 28
  The amelioration of the wound bed conditions will be evaluated:
  - by measuring the proportion of patients having an increase of at least one subclass of the WBS (0-16 score; 0 worse score-16 best score possible) from baseline to 7, 21 and 28 days of treatment with ConnettivinaBio Plus cream compared to ConnettivinaBio cream;
improving the wound bed condition | At days 7, 14, 21 and 28
  The amelioration of the wound bed conditions will be evaluated:
  - by measuring the percentage change from baseline in the WBS (0-16 score; 0 worse score-16 best score possible) after 7, 14, 21, and 28 days of treatment with ConnettivinaBio Plus cream compared to ConnettivinaBio cream.
control of bacterial load of wounds | At days 7, 14, 21 and 28
  The performance of ConnettivinaBio Plus in the bacterial load control will be evaluated by measuring the change from baseline of CFU/ml derived from the culture of a swab collected according to the Levin's technique, after 7, 14 and 28 days of treatment and compared to ConnettivinaBio cream
control on signs of wound infection | At days 7, 14, 21 and 28
  Difference in the performance of ConnettivinaBio Plus, compared to ConnettivinaBio, with respect to clinical signs of wound infection. The appearance and/or modification of signs of infection will be evaluated as percentage change from baseline at all visits. The evaluation will be carried out calculating the clinical wound's infection score through an 18-point scale, based on the presence and intensity of the following clinical signs: fever, local heat, peri-lesional erythema, persistent pain (between two dressing changes), oedema, malodour, pus and exudate production (Cutting KF, 1994; Trial C, 2010).
improving the reepithelization rate | At days 7, 21 and 28
  The reepithelization rate will be evaluated as the difference in the mean percentage reduction of lesion area from baseline between patients treated with ConnettivinaBio Plus versus ConnettivinaBio at all the visits by using a computerized image software (Chang AC, 2011) and as a distribution of percentage reduction in the following classes: ≤25%; >25% and ≤50%; >50% and ≤75%; >75% and ≤95%; >95% and ≤100% of the lesion area.
improving patient's quality of life | At days 7, 14, 21 and 28
  Patient's quality of life assessment will be evaluated as a change from baseline after 7, 14, 21 and 28 days, through administration of EuroQoL-5D (EQ-5D)
clinician's global assessment of the lesion | At days 7, 14, 21 and 28
  Clinical Global Assessment (CGA) will be evaluated at each post baseline visit: the clinician will be requested to score the lesion on a five grade scale: 1= worsening, 2= no change, 3= minimal improvement, 4= moderate improvement and 5= good improvement
easiness of the treatment application | at day 28
  The easiness of the treatment application will be appraised by the Un-blinded Investigator and by the patient after 28 days as excellent, good, acceptable, bad or unacceptable.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | throughout study completion, an average of 1 year
  The safety and tolerability of treatment will be assessed by investigating local and expected adverse events, as consequence of the product application and any other adverse event occurred during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Casa di Cura Villa Donatello, Florence, Italy